CLINICAL TRIAL: NCT07205185
Title: A Multicenter, Single-arm, Prospective Phase II Clinical Study of Epalrotokewali Monotherapy Combined With Eribulin, Anlotinib, and Radiotherapy for the Treatment of Patients With Advanced Soft Tissue Sarcoma.
Brief Title: A Multicenter, Single-arm, Prospective Phase II Clinical Study of Epalrotokewali Combined With Eribulin, Anlotinib, and Radiotherapy for the Treatment of Patients With Advanced Soft Tissue Sarcoma.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RITEA
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Soft Tissue Sarcoma (STS)
MeSH Terms: conditions — Sarcoma | interventions — eribulin; anlotinib; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706+ Eribulin + Anlotinib + Radiotherapy (Experimental): QL1706:5 mg/kg, intravenous injection (IV) on Day 1, every 3 weeks (Q3W). Eribulin : 1.1 mg/m², intravenous infusion (IV) on Days 1 and 8, Q3W. Anlotinib : Oral administration before breakfast, 12 mg once daily (QD) on Days 1-14, followed by a 1-week drug holiday, Q3W.
  Radiotherapy : Hypofractionated radiotherapy, 15-60 Gy delivered in 5-8 fractions.
  Interventions: Drug: QL1706 + Eribulin + Anlotinib + Radiotherapy

INTERVENTIONS:
Drug: QL1706 + Eribulin + Anlotinib + Radiotherapy — QL1706: 5 mg/kg, intravenous injection (IV) on Day 1, every 3 weeks (Q3W). Eribulin : 1.1 mg/m², intravenous infusion (IV) on Days 1 and 8, Q3W. Anlotinib : Oral administration before breakfast, 12 mg once daily (QD) on Days 1-14, followed by a 1-week drug holiday, Q3W.
  Radiotherapy : Hypofractionated radiotherapy, 15-60 Gy delivered in 5-8 fractions.
  Eribulin is administered for 6 cycles. Epalizumab and anlotinib are continued until disease progression, intolerable toxicity, initiation of new anti-tumor treatment, loss to follow-up, death, or withdrawal from the study (whichever occurs first).

SUMMARY:
This study intends to enroll patients with advanced soft tissue sarcoma, employing immunotherapy combined with eribulin, anlotinib, and radiotherapy as subsequent-line treatment to preliminarily explore its efficacy and safety. QL1706, a dual-targeting agent against PD-1 and CTLA-4, has been approved by the National Medical Products Administration (NMPA) of China for the second-line treatment of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Subjects aged 14-75 years;
* Patients with histologically or cytologically confirmed advanced soft tissue sarcoma (STS);
* Patients with STS who have failed first-line or higher treatment;
* At least one measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1);
* ECOG performance status (PS) score of 0-1;
* Adequate organ and bone marrow function, with laboratory tests meeting the following criteria within 7 days prior to the first dose of study drug (without having received any blood components, hematopoietic growth factors, albumin, or other medications considered corrective therapy by the investigator within 14 days prior to testing):

  i. Hematology: Hemoglobin (Hb) ≥90 g/L, absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count (PLT) ≥90×10⁹/L.

ii. Biochemistry: Serum creatinine (Cr) ≤1.5×upper limit of normal (ULN); serum total bilirubin (TBIL) ≤1.5×ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0×ULN for subjects without liver metastases, and ALT and AST ≤5.0×ULN for subjects with liver metastases; serum albumin (ALB) ≥25 g/L.

iii. Coagulation function: International normalized ratio (INR) ≤1.5×ULN; prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN (for subjects receiving prophylactic anticoagulation therapy, the investigator should assess that INR and APTT are within safe and effective therapeutic ranges);

* Women of childbearing potential must use reliable contraception from screening until 3 months after discontinuation of trial medication, and have a negative pregnancy test (serum or urine) within 7 days prior to enrollment. Men must agree to use appropriate contraception or have undergone surgical sterilization from screening until 3 months after discontinuation of trial medication;
* Expected survival time ≥12 weeks.

Exclusion Criteria:

* History of allergy to QL1706 or any of its components, or contraindication to its treatment;
* Prior administration of QL1706 or eribulin;
* Specific pathological subtypes, such as Ewing sarcoma, non-poly-morphic rhabdomyosarcoma, or gastrointestinal stromal tumor (GIST);
* Resistance or intolerance to anlotinib, eribulin, radiotherapy, or any other contraindications to these treatments;
* Use of any other investigational drug within 4 weeks prior to screening or participation in another clinical trial;
* Diagnosis of immunodeficiency or ongoing systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first trial treatment;
* Known history of active Mycobacterium tuberculosis (TB) infection;
* Known history of human immunodeficiency virus (HIV) infection;
* Active brain metastases or meningeal metastases;
* Uncontrolled hypertension (systolic blood pressure [SBP] ≥140 mmHg or diastolic blood pressure [DBP] >90 mmHg despite optimal medical therapy);
* Severe cardiovascular disease: myocardial ischemia of grade II or higher, myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥450 ms in males or ≥470 ms in females); NYHA class III-IV heart failure, or left ventricular ejection fraction (LVEF) <50% as assessed by echocardiography;
* Respiratory syndrome (dyspnea of CTCAE grade ≥2), or uncontrolled serous cavity effusion (including pleural effusion, ascites, or pericardial effusion);
* Active hepatitis C and/or hepatitis B infection (hepatitis B: HBsAg-positive with HBV DNA ≥500 IU/mL; hepatitis C: HCV RNA-positive);
* Major surgical procedure, severe traumatic injury, fracture, or ulcer within 4 weeks prior to randomization;
* History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), inflammatory bowel disease (IBD), vascular thrombosis associated with antiphospholipid syndrome (APS), Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome (GBS), multiple sclerosis (MS), vasculitis, or glomerulonephritis;
* Medical history, diseases, treatments, or laboratory abnormalities that may interfere with trial results, prevent the subject from completing the study, or other conditions deemed unsuitable for study participation by the investigator.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  The percentage of subjects achieving complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
DCR | up to two years
  The percentage of subjects achieving complete response (CR), partial response (PR), or stable disease (SD).
PFS | up to two years
  From the date of enrollment, the date of the first documented tumor progression (assessed by RECIST v1.1 criteria, regardless of whether treatment is continued) or the date of death from any cause, whichever occurs first.
OS | up to two years
  The time from the initiation of treatment to death from any cause in subjects.
6-month PFS rate | up to six months
  The percentage of patients with no progression at 6 months of treatment.
DoR | up to two years
  For patients who achieved complete response (CR) or partial response (PR), the time from the first tumor assessment documenting response to disease progression or death, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No